CLINICAL TRIAL: NCT03118830
Title: Long Protocol and Freeze All Embryos vs Antagonist Protocol With Fresh Embryo Transfer in PCOS Patients Undergoing ICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 164
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Triptorelin Pamoate; cetrorelix; Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long GnRH agonist (Active Comparator): daily SC injection of Triptorelin :Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l with either HMG or rFSH in a starting dose of 150-300 IU/day
  Interventions: Drug: Triptorelin; Drug: Recombinant Follicle Stimulating Hormone
- GnRH antagonist (Active Comparator): Flexible GnRH antagonist protocol was done with daily s.c administration of cetrorelix 0.25 mg started when one or more of the following criteria were achieved: (i) one or more follicle reached 14 mm diameter; (ii) The level of serum E2 reached 600 pg/ml; and (iii) The level of serum LH levels reached 10 IU/l. Daily sc rFSH injections was started on 2nd day of the cycle in the antagonist protocol. Continuation of rFSH and GnRH antagonist daily until triggering day was done
  Interventions: Drug: cetrorelix; Drug: Recombinant Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Triptorelin — daily SC injection of Triptorelin 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering.
  Other Names: Decapeptyl
  Arms: Long GnRH agonist
Drug: cetrorelix — Flexible GnRH antagonist protocol was done with daily s.c administration of cetrorelix 0.25 mg started when one or more of the following criteria were achieved: (i) one or more follicle reached 14 mm diameter; (ii) The level of serum E2 reached 600 pg/ml; and (iii) The level of serum LH levels reached 10 IU/l .
  Other Names: Cetrotide
  Arms: GnRH antagonist
Drug: Recombinant Follicle Stimulating Hormone — Daily sc rFSH (Gonal-f; Merck Serono , Darmstadt, Germany) injections was started on 2nd day of the cycle in the antagonist protocol. Continuation of rFSH and GnRH antagonist daily until triggering day was done.
  Other Names: Gonal-f

SUMMARY:
Patients will be divided into two groups Group A; patients using long protocol and freeze all embryos Group B; patients using antagonist protocol with fresh embryo transfer Patients will be carefully chosen according to a strict inclusion and exclusion criteria after meticulous revision of patient files.

In the long protocol, daily SC injection of Triptorelin :Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day according to women age, day 3 FSH,AMH and previous gonadotropin response then adjustment of the dose according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day (6) for folliculometry and endometrial thickness and pattern.

Triggering by HCG 10000 IU IM (Pregnyl, Organon, the Netherlands) when 2 or more follicles have 18 mm as a mean diameter .

Flexible GnRH antagonist protocol was done with daily s.c administration of cetrorelix 0.25 mg (Cetrotide, Merck Serono, Darmstadt, Germany) started when one or more of the following criteria were achieved: (i) one or more follicle reached 14 mm diameter; (ii) The level of serum E2 reached 600 pg/ml; and (iii) The level of serum LH levels reached 10 IU/l . Daily sc rFSH (Gonal-f; Merck Serono , Darmstadt, Germany) injections was started on 2nd day of the cycle in the antagonist protocol. Continuation of rFSH and GnRH antagonist daily until triggering day was done.

DETAILED DESCRIPTION:
Patients will be divided into two groups Group A; patients using long protocol and freeze all embryos Group B; patients using antagonist protocol with fresh embryo transfer Patients will be carefully chosen according to a strict inclusion and exclusion criteria after meticulous revision of patient files.

In the long protocol, daily SC injection of Triptorelin :Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG triggering. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day according to women age, day 3 FSH,AMH and previous gonadotropin response then adjustment of the dose according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day (6) for folliculometry and endometrial thickness and pattern.

Triggering by HCG 10000 IU IM (Pregnyl, Organon, the Netherlands) when 2 or more follicles have 18 mm as a mean diameter .

Flexible GnRH antagonist protocol was done with daily s.c administration of cetrorelix 0.25 mg (Cetrotide, Merck Serono, Darmstadt, Germany) started when one or more of the following criteria were achieved: (i) one or more follicle reached 14 mm diameter; (ii) The level of serum E2 reached 600 pg/ml; and (iii) The level of serum LH levels reached 10 IU/l . Daily sc rFSH (Gonal-f; Merck Serono , Darmstadt, Germany) injections was started on 2nd day of the cycle in the antagonist protocol. Continuation of rFSH and GnRH antagonist daily until triggering day was done.

Cycle cancellation was decided when transvaginal ultrasound scan on cycle day (9) revealed no adequate follicular growth (<3 mature follicles),if no oocytes were retrieved on ovum pick up,or if failure of fertilization occurred. If signs of early OHSS were observed at 3rd day of ovum pickup ,cancellation of ET was done with elective embryo cryopreservation as it may end with life-threatening OHSS . ET was cancelled also if any criteria of hospital admission was found

ELIGIBILITY:
Inclusion Criteria:

1. PCOS diagnosed by Roterdam criteria
2. Protocol used for ovulation induction either long procol with freeze all embryos vs antagonist with fresh embryo transfer
3. BMI less than 30
4. ALL patients receiving adjuvant drugs for prevention of OHSS in the form of metformin, cabergoline as well as prophylactic hysteril , low dose asprin and LMW heparin following oocyte retrieval on a routine basis

Exclusion criteria;

1. PCOS on long protocol with fresh embryo transfer and those on antagonist protocol with freezing all embryo
2. BMI more than 30
3. PCOS patients not given adjuvant drugs in prophylaxis of OHSS
4. Antagonist cases receiving agonist as trigger instead of HCG
5. PCOS receiving more than 5000 IU HCG as trigger
6. PCOS undergoing costing during ovulation induction
7. PCOS with known medial problems as diabetes or hypertension

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 204 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  The detection of fetal cardiac activity within a gestational sac on ultrasonography examinationenlargement (<12 cm in average diameter), ascitis in moderate form and clinical evidence of ascites and/or hydrothorax, haemoconcentration and significant ovarian enlargement (>12 cm in average diameter)

SECONDARY OUTCOMES:
chemical pregnancy rate | 14 days after embryo transfer
  POSITIVE pregnancy testing of HCG exceeding 50 mIU
abortion rate | 12 weeks of gestational age
  termination of pregnancy before 12 weeks of gestational age
Ovarian hyperstimulation syndrome | 7 days after HCG administration
  evaluated by the British fertility society criteria, the Canadian Fertility and Andrology Society ( CFAS) and the Society of obstetrics and Gynecology of Canada (SOGC); [Mild OHSS; Abdominal bloating, Mild abdominal pain, Ovarian size usually < 8 cm. Moderate OHSS; Moderate abdominal pain, Nausea with/without vomiting, Ultrasound evidence of ascites and Ovarian size usually 8-12 cm. Severe OHSS; Clinical ascites (occasionally pleural effusion), Oliguria, Hemoconcentration with hematocrit (> 45%), Hypoproteinemia and Ovarian size usually > 12 cm. Critical OHSS; Tense ascites or large pleural effusion, Hematocrit (> 55%) White cell count > 25 000/L, anuria, Thromboembolism or Acute respiratory distress syndrome
Late Ovarian hyperstimulation syndrome | 12 to 17 days following HCG administration
  OHSS manifestation 12 to 17 days following HCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Ahmed Maged, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes